CLINICAL TRIAL: NCT05533580
Title: Differential Effects of Remimazolam and Propofol on Dynamic Cerebral
Brief Title: Differential Effects of Remimazolam and Propofol on Dynamic Cerebral Autoregulation During General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Fuzhou Hua, Chief Physician, Second Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-TCD-1
Record Dates: First submitted 2022-09-02; First posted 2022-09-09 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: General Anesthesia; Laparoscopic Cholecystectomy; Remimazolam; Propofol; Dynamic Cerebral Autoregulation
Keywords: General Anesthesia; Laparoscopic Cholecystectomy; Remimazolam; Propofol; dynamic cerebral autoregulation
MeSH Terms: interventions — remimazolam; Sufentanil; cisatracurium; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): 1. Induction of anesthesia Slowly injects remimazolam 0.4-0.6 mg/kg (about 1 minute) until loss of consciousness (LoC), if the degree of sedation is insufficient, additional remimazolam (0.05 mg/kg each time) is allowed. After the LoC, intravenous sufentanil 0.3 ~0.5ug/kg and cisatracurium besylate 0.1 mg/kg are injected intravenously. After the muscles are sufficiently relaxed and blood circulation is stable, the tracheal tube is inserted under a glide scope.
  2. Maintenance of anesthesia remimazolam 0.4~1.2 mg/kg/h and remifentanil 0.1~0.3 ug/kg/min are injected intravenously to maintain sedation and assistant analgesia, and cisatracurium besylate 0.02 mg/kg is allowed to add as appropriate. During the operation, the dose of anesthetic drugs is adjusted so that the fluctuation of heart rate and blood pressure did not exceed 10 %.
  Interventions: Drug: Remimazolam
- Propofol group (Active Comparator): 1. Induction of anesthesia Slowly injects propofol 2-4 mg/kg (about 1 min) until loss of consciousness (LoC), allowing additional propofol (0.5 mg/kg each time) if sedation is insufficient. after LoC, intravenous sufentanil 0.3 ~0.5ug/kg and cisatracurium besylate 0.1 mg/kg. after sufficient muscle relaxation and blood circulation stabilization, the tracheal tube was inserted under the sliding scope.
  2. Maintenance of anesthesia propofol 4~10mg/kg/h and remifentanil 0.1~0.3 ug/kg/min are injected intravenously to maintain sedation and assistant analgesia, and cisatracurium besylate 0.02 mg/kg is allowed to add as appropriate. During the operation, the dose of anesthetic drugs is adjusted so that the fluctuation of heart rate and blood pressure did not exceed 10 %.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — The experimental group was sedated with remimazolam.
  Other Names: sufentanil; cisatracurium besylate
  Arms: Remimazolam group
Drug: Propofol — The control group was sedated with propofol.
  Other Names: sufentanil; cisatracurium besylate
  Arms: Propofol group

SUMMARY:
Cerebral autoregulation (CA) is the property of the cerebral vascular bed to maintain cerebral perfusion in the presence of changes in blood pressure. In the case of anesthesia, altered cerebral autoregulation, including altered carbon dioxide and hemodilution, can impair physiological changes in the body and lead to poor postoperative prognosis. As a novel ultra-short-acting benzodiazepines drugs, remimazolam has been accepted for induction and maintenance of clinical anesthesia. Compared to the traditional benzodiazepines drugs, remimazolam combines the safety of midazolam with the effectiveness of propofol, and also has the advantages of acting quickly, short half-life, no injection pain, slight respiratory depression, independent of liver and kidney metabolism, long-term infusion without accumulation, and has a specific antagonist: flumazenil. Our study aimed to investigate the different effects of remimazolam and propofol on dynamic cerebral blood flow autoregulation function during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years, gender not limited
2. Patients proposed to undergo elective laparoscopic cholecystectomy under general anesthesia, with an expected operative length of approximately 1h~2h
3. Good penetration of the temporal window.
4. ASA anesthesia classification grade I to II.
5. can communicate effectively with the physician.
6. Patients were aware of and voluntarily signed the informed consent form.

Exclusion Criteria:

1. Relative contraindications to general anesthesia: patients with severe heart and lung function diseases.
2. History of syncope, and dizziness.
3. Patients with a history of psychiatric disorders, neurological disorders, drug abuse, or drug addiction
4. Patients with cerebrovascular or carotid artery lesions;
5. Those who are unable to cooperate in completing the test
6. Persons who have taken benzodiazepines intermittently in the last three months.
7. Those with known allergies or allergies to the test drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Differences in dynamic cerebral blood flow autoregulation | From the time the patient enters the operating room to the time they leave the operating room, one and a half hours on average.
  Comparison of the consistency, gain and phase of the transfer function parameters in the frequency range of 0.02-0.07 Hz, 0.07-0.2 Hz and 0.2-0.5 Hz for the propofol and rimazolam groups, respectively.

SECONDARY OUTCOMES:
systolic pressure | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
diastolic pressure | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
mean pressure | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
heart rate | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
pulse | Up to 5 hours including preoperative, intraoperative, and postoperative periods
  Indicators related to perioperative hemodynamics
Recovery times | Up to 30 minutes after operation
  The period from discontinuation of anesthetic drugs to the recovery of the patient's self-consciousness and can respond correctly to external stimuli. All the patients can be allowed to leave the post-anesthesia care unit after Aldrete ≥ 9. Delayed awakening is defined as failure to achieve Aldrete ≥ 9 more than 30 minutes after surgery.
Complication | During the perioperative period
  All the perioperative complications are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Nanchang University, Nanchang University, Nanchang, Jiangxi, China